CLINICAL TRIAL: NCT00119548
Title: Improving HIV Screening by Nurse Rapid Testing, Streamlined Counseling
Brief Title: Improving HIV Screening With Nurse-Based Rapid Testing/Streamlined Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IIR 04-023; PCC 2004-081171; NCT00186160 (obsolete NCT alias)
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Health Care Quality, Access, and Evaluation; Delivery of Health Care; Immune System Diseases; HIV Infections
Keywords: HIV Rapid Testing; Cost-effectiveness; HIV Seronegativity
MeSH Terms: conditions — Immune System Diseases; HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Other): Randomized, controlled trial with three intervention models: Model A (traditional counseling/testing);
  Interventions: Other: Rates of HIV testing and receipt of results; Other: Sexual risk reduction; HIV knowledge improvement
- Arm 2 (Other): Model B (nurse-initiated screening, traditional counseling/testing);
  Interventions: Other: Rates of HIV testing and receipt of results; Other: Sexual risk reduction; HIV knowledge improvement
- Arm 3 (Other): Model C (nurse-initiated screening, streamlined counseling/rapid testing).
  Interventions: Other: Rates of HIV testing and receipt of results; Other: Sexual risk reduction; HIV knowledge improvement

INTERVENTIONS:
Other: Rates of HIV testing and receipt of results — Rates of HIV testing and receipt of results
  Arms: Arm 1
Other: Sexual risk reduction; HIV knowledge improvement — Sexual risk reduction; HIV knowledge improvement
  Arms: Arm 1
Other: Rates of HIV testing and receipt of results — Rates of HIV testing and receipt of results
  Arms: Arm 2
Other: Sexual risk reduction; HIV knowledge improvement — Sexual risk reduction; HIV knowledge improvement
  Arms: Arm 2
Other: Rates of HIV testing and receipt of results — Rates of HIV testing and receipt of results
  Arms: Arm 3
Other: Sexual risk reduction; HIV knowledge improvement — Sexual risk reduction; HIV knowledge improvement
  Arms: Arm 3

SUMMARY:
Background: HIV testing is cost-effective in unselected general medical populations, yet testing rates among those at-risk remain low, even among those with regular primary care. HIV rapid testing is effective in many healthcare settings but scant research has been done within primary care settings, nor within the US Department of Veteran's Affairs Healthcare System.

Objectives: We evaluated three methods proven effective in other diseases/settings: Nurse standing orders for testing, streamlined counseling, and HIV rapid testing.

Design: Randomized, controlled trial with three intervention models: Model A (traditional counseling/testing); Model B (nurse-initiated screening, traditional counseling/testing); Model C (nurse-initiated screening, streamlined counseling/rapid testing).

Participants: 251 patients with primary/urgent care appointments in two VA clinics in the same city (one large urban hospital, one freestanding outpatient clinic in a high HIV prevalence area)

Measurements: Rates of HIV testing and receipt of results; sexual risk reduction; HIV knowledge improvement.

Results: Testing rates were 40.2% (Model A), 84.5% (Model B), and 89.3% (Model C) (p=<.01). Test receipt rates were 14.6% (Model A), 31.0% (Model B), 79.8% (Model C) (all p=<.01). Sexual risk reduction and knowledge improvement did not differ significantly between counseling methods.

Conclusions: Streamlined counseling with rapid testing significantly increased testing and receipt rates over current practice without changes in risk behavior or post-test knowledge. Increased testing and receipt of results could lead to earlier disease identification, increased treatment and reduced morbidity/mortality. Policymakers should consider streamlined counseling/rapid testing when implementing routine HIV testing into primary/urgent care.

DETAILED DESCRIPTION:
BACKGROUND/RATIONALE:

HIV testing is cost-effective in unselected general medical populations, yet testing rates among those at-risk remain low, even among those with regular primary care. HIV rapid testing is effective in many healthcare settings but scant research has been done within primary care settings, nor within the US Department of Veteran's Affairs Healthcare System.

The cumbersome nature and complexity of current counseling and testing procedures have been suggested as reasons that rates of receipt of HIV test results are so low. Because the standard screening test results are unavailable on the same day, many persons do not return for the results. Up to 30% of persons who tested HIV-positive during 2000 and 39% of persons who tested HIV-negative did not return (1). The CDC has recommended that alternate streamlined counseling and testing methods may increase the receipt rates of HIV tests. To address the problems of failing to return for screening results, we incorporated rapid HIV testing into the proposed screening trial.

OBJECTIVE(S):

The specific aims of this project were:

To determine whether nurse-based referral for traditional HIV testing and counseling will improve screening rates compared to current testing procedures.

To determine whether nurse-based rapid testing with streamlined counseling improves screening rates more than nurse-based referral for traditional testing and counseling alone.

To assess the cost-effectiveness of these alternative strategies for HIV testing and counseling.

Secondary aims were to compare patient knowledge of HIV testing prevention practices and their views of the procedures' acceptability after traditional and rapid testing/streamlined counseling. To achieve these aims, we proposed a robust three-arm randomized controlled trial.

METHODS:

We planned a parallel-group randomized controlled trial set in the general medicine and urgent care clinics of the West Los Angeles VA Medical Center (VAMC). All participants underwent an interview collecting information about HIV risk factors and other predictors of HIV screening, as well as knowledge of HIV test characteristics and prevention. All patients were randomized to one of three models of screening: Model A: Traditional counseling/testing; Model B: Nurse-based screening + traditional counseling/testing; Model C: Nurse-based screening + streamlined counseling/ rapid testing

The analysis focused on differences between the three models in rates of screening, receipt of results, knowledge, acceptability and cost-effectiveness.

FINDINGS/RESULTS:

Testing rates were 40.2% (Model A), 84.5% (Model B), and 89.3% (Model C) (p=<.01). Rates of receipt of test results were 14.6% (Model A), 31.0% (Model B), 79.8% (Model C) (all p=<.01). Reduction in sexual risk and HIV knowledge improvement did not differ significantly between traditional versus streamlined counseling.

IMPACT:

Streamlined counseling with rapid testing significantly increased testing and receipt rates over current practice without changes in risk behavior or post-test knowledge. Increased testing and receipt of results could lead to earlier disease identification, increased treatment and reduced morbidity/mortality. Policymakers should consider streamlined counseling/rapid testing when implementing routine HIV testing into primary/urgent care.

Widespread implementation would lead to critically important health benefits for veterans: 1) Increased rates of testing, which would lead to earlier identification of disease, increased treatment and decreased HIV transmission, morbidity and mortality; 2) Lower screening costs without decrements in either patient knowledge or acceptability.

The CDC has made identification of people with HIV a national priority. The VA has an opportunity to provide national leadership in elucidating how best to identify people living with HIV and ensure access to state-of-the-art care.

ELIGIBILITY:
Inclusion Criteria:

Seeing a provider the day of recruitment Between 18-65 years of age Unaware of HIV status Has not had an HIV test in past year Able to communicate fluently in English Competent to consent to participation and HIV testing

Exclusion Criteria:

Not between 18-65 yrs. of age aware of HIV status has had HIV test within past year cannot communicate in English deemed incompetent to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To determine whether nurse-based referral for traditional HIV testing and counseling will improve screening rates compared to current testing procedures.To determine whether nurse-based rapid testing with streamlined counseling improves screening rates | 90 days

SECONDARY OUTCOMES:
To compare patient knowledge of HIV testing prevention practices and their views of the procedures' acceptability after traditional and rapid testing/streamlined counseling. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Asch, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Douglas K. Owens, MD MS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Result] Pinkerton SD, Bogart LM, Howerton D, Snyder S, Becker K, Asch SM. Cost of OraQuick oral fluid rapid HIV testing at 35 community clinics and community-based organizations in the USA. AIDS Care. 2009 Sep;21(9):1157-62. doi: 10.1080/09540120902729940. PMID 20024775
- [Result] Anaya HD, Hoang T, Golden JF, Goetz MB, Gifford A, Bowman C, Osborn T, Owens DK, Sanders GD, Asch SM. Improving HIV screening and receipt of results by nurse-initiated streamlined counseling and rapid testing. J Gen Intern Med. 2008 Jun;23(6):800-7. doi: 10.1007/s11606-008-0617-x. Epub 2008 Apr 18. PMID 18421508